CLINICAL TRIAL: NCT00057798
Title: Molecular And Genetic Changes In Patients With Resectable Non-Small Cell Lung Cancer (NSCLC) Following Neoadjuvant Chemotherapy With Vinorelbine And Gemcitabine - Phase II Study
Brief Title: Genetic Changes in Patients With Non-Small Cell Lung Cancer Who Are Receiving Vinorelbine and Gemcitabine Before Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Nithya Ramnath, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000270753; RPCI-RP-00-01
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Vinorelbine; Cytogenetic Analysis; Microarray Analysis; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: vinorelbine ditartrate
Genetic: cytogenetic analysis
Genetic: loss of heterozygosity analysis
Genetic: microarray analysis
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Determination of genetic changes in patients with non-small cell lung cancer may help predict the outcome of treatment. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them before surgery, may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study genetic changes and the effectiveness of combining vinorelbine with gemcitabine before surgery in treating patients who have stage IB, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of expression of epithelial markers CK19, CK20, MUC1, and MUC5 (by reverse transcriptase-polymerase chain reaction) in lymph node tissue and blood samples of patients with resectable stage IB-III non-small cell lung cancer treated with neoadjuvant vinorelbine and gemcitabine followed by surgery.
* Determine the expression of the multidrug resistance-associated protein gene before and after treatment with this regimen in these patients.
* Determine the global expression profile of genes (by microarray technology) in tumor tissue of patients treated with this regimen.
* Determine the frequency of loss of heterozygosity at several loci on chromosomes 3p, 9p, and 11p before and after treatment with this regimen in these patients.
* Determine the percent positivity of cells that stain for MCM2 and CDC6 (prereplicative complex) by immunohistochemistry before and after treatment with this regimen in these patients.
* Determine the feasibility of this regimen in these patients.
* Determine the pathological response rates in patients treated with this regimen.
* Determine the side effects of this regimen in these patients.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Determine the autologous immune response in patients treated with this regimen.

OUTLINE: Patients receive vinorelbine IV over 6-10 minutes and gemcitabine IV over 30 minutes on days 1, 8, 22, and 29 in the absence of disease progression or unacceptable toxicity.

Patients with no disease progression by scans or bronchoscopy undergo surgical resection between days 57-70 (weeks 8-10).

Loss of heterozygosity (LOH) at loci on chromosomes 3p, 9p, and 11p is assessed in blood specimens, tumor tissue, and noncancerous tissue before and after chemotherapy. Specimens are also examined for molecular markers of occult metastasis using reverse transcriptase-polymerase chain reaction. Multidrug resistance-associated protein gene expression is also determined using microarray technology.

Patients are followed every 3 months for 2 years, every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell carcinoma of the lung

  * May be confirmed at the initial bronchoscopy and mediastinoscopy
  * Stage IB (T2, N0, M0)
  * Stage IIA (T1, N1, M0)
  * Stage IIB (T2-3, N0-1, M0)
  * Stage IIIA (T1-3, N1-2, M0)
  * stage IIIB (2 lesions in 1 lobe [T4])
* No N3 lymph nodes (contralateral mediastinal/hilar and supraclavicular/scaline) OR T4 primary tumor (malignant pleural effusion or mediastinal invasion) by clinical staging criteria (seen on CT or PET scan and proven by mediastinoscopy)
* No metastatic disease (except N1 or N2 disease) or malignant pleural effusion* detected on preoperative evaluation

  * No exudative effusions (even if cytologically negative)

    * Pleural fluid is considered exudative if the following apply:

      * Ratio of pleural fluid protein to serum protein is greater than 0.5
      * Ratio of pleural fluid lactic dehydrogenase (LDH) to serum LDH is at least 0.6
      * Pleural fluid LDH is greater than 200 IU/L
  * No multiple areas of fluorodeoxyglucose (FDG) uptake** outside the area of the primary tumor in the lung NOTE: *Effusions visible only on CT scan and not large enough for safe thoracentesis are allowed

NOTE: **If only 1 area shows an increase in FDG uptake, the area of concern requires further evaluation (e.g., biopsy) to exclude metastatic disease

* Bidimensionally measurable or evaluable disease* NOTE: *Lesions apparent on chest CT scan (e.g., ill-defined masses associated with post obstructive changes and mediastinal or hilar adenopathy measurable in 1 dimension) are considered evaluable

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST or ALT no greater than 1.5 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Deemed medically fit for surgical resection
* No other active malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No psychological, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent participation in the RPCI vaccine study (postoperative vaccination with autologous tumor-associated antigen-pulsed dendritic cells) is allowed

Chemotherapy

* No prior chemotherapy for lung cancer
* No concurrent participation in another study involving other chemotherapy agents

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for lung cancer
* No concurrent participation in another study involving radiotherapy

Surgery

* No prior surgery for lung cancer
* More than 3 months since other prior major surgery (e.g., coronary artery bypass graft)

Other

* No other prior therapy for lung cancer
* No other concurrent antineoplastic agents
* Concurrent participation in observational studies requiring bloodwork, radiographs, pulmonary function tests, or quality of life studies is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-03; Primary Completion 2003-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Ramnath N, Sommers E, Anderson T, et al.: Neoadjuvant gemcitabine and vinorelbine in non-small-cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2818, 2003.